CLINICAL TRIAL: NCT01473121
Title: Profile of the Hepatocellular Carcinoma Patients in Turkey
Brief Title: Hepatocellular Carcinoma Registry for Turkey (3K Trial)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15807; NX1110TR (Other: company internal)
Record Dates: First submitted 2011-11-02; First posted 2011-11-17 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Registry; Turkey
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — All treatment options (inc. surgery, TACE, drugs) will be registered.

SUMMARY:
This registry study is national, multi-center, prospective study without any interventions to the treatment strategies and/or decisions of the investigators. It is designed in order to determine the general profile of HCC patients in Turkey. Socio-demographic characteristics, family history, medical history and treatment pattern of HCC patients will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with hepatocellular carcinoma in last 3 months
* To be older than 18 years old
* To sign informed consent form (ICF)

Exclusion Criteria:

* Patients that does not sign or withdraw informed consent form.
* According to investigator's opinion; existence of any situation/condition that will significantly complicate patient follow up.
* Currently or previously taking part in 3K observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are diagnosed with hepatocellular carcinoma in last 3 months
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2012-08-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Descriptive analysis of HCC risk factors | Baseline
  i.e. smoking and alcohol consumption status; family history for hepatitis, HCC, and other malignancies; history of hepatic disease and blood transfusion; concomitant diseases; treatments applied
Descriptive analysis of clinical profile of newly diagnosed HCC patients | Baseline

SECONDARY OUTCOMES:
Number of participants with underlying liver disease and family history | Baseline
Treatment options as applied by doctors to HCC patients | Up to approximately 5 years
Overall survival time since diagnosis | Up to approximately 5 years
Number of participants with adverse events | Up to approximately 5 years
Descriptive analysis of demographic characteristics of HCC patients | Baseline
Descriptive analysis of clinical characteristics of HCC patients | Up to approximately 5 years
Descriptive analysis of tumor properties | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Turkey (Türkiye)